CLINICAL TRIAL: NCT00713895
Title: Treating Chinese Smokers With Interactive Expert System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Janice Tsoh, Ph.D., Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5K23DA000468 (NIH); 5K23DA000468 (NIH)
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; randomized trial; Asian; Chinese American; stages of change
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Self-Help (Active Comparator): receive a standard self-help manual in Chinese and English of the participants' choice at baseline
  Interventions: Behavioral: Standard Self-Help
- Expert System (Experimental): receive an expert system intervention that included the Pathway-To-Change self-help manual and a series of 3 individualized feedback reports at baseline, 3, and 6 months.
  Interventions: Behavioral: Expert System

INTERVENTIONS:
Behavioral: Expert System — an expert system intervention provided the Pathway-To-Change self-help manual and a series of 3 individualized feedback reports at baseline, 3, and 6 months.
  Arms: Expert System
Behavioral: Standard Self-Help — standard smoking cessation self-help manual
  Arms: Standard Self-Help

SUMMARY:
The research study examined the feasibility, implementation, and efficacy of the interactive expert system intervention for smoking cessation in the Chinese American population.

DETAILED DESCRIPTION:
The research study examines the feasibility, implementation, and efficacy of the interactive expert system intervention for smoking cessation in the Chinese American population. The primary specific aim of the proposed research is to test the following hypotheses: 1) Proactive recruitment approach will be more effective in recruiting smokers who are in precontemplation (no intent to quit smoking in the next 6 months) than a reactive approach. 2) Participants in the experimental condition receiving the interactive stage-matched expert system intervention plus a manual will be more likely to be abstinent at 12 and 18 than those in the control condition receiving a non-interactive standard manual. 3) Participants receiving the interactive expert system intervention will be more likely to report at least one quit attempt than those in the control condition at months 6, 12, and 18. 4) Participants receiving the interactive expert system intervention will be more likely to have a significant decrease in number of cigarettes smoked than those in the control condition at months 3, 6, 12, and 18. After the intervention adaptation and the pilot testing phase of study procedures, the study will achieve the above aims using a randomized trial targeting 400 Chinese American Smokers with follow-up assessments at 3, 6, 12, and 18 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* residents of the San Francisco Bay Area
* age 18 or older
* self-identified as Chinese in ethnicity
* able to read English or Chinese
* have smoked at least 100 cigarettes in their lifetime
* currently smoke at least 5 cigarettes in the past 7 days

Exclusion Criteria:

* currently engaging in other smoking cessation efforts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2001-08; Primary Completion 2004-01 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
abstinence | 18 months
  self-report 7-day point prevalence abstinence of cigarette use

SECONDARY OUTCOMES:
quit attempt | 18 months
  self-report of 24-hour quit attempt
reduction | 18 months
  smoking reduction from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Janice Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Langley Porter, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No